CLINICAL TRIAL: NCT06341270
Title: Efficacy of Transcutaneous Electrical Acupoint Stimulation on Postoperative Pain and Recovery in Patients Undergoing Hepatectomy：a Prospective, Randomized Controlled Trial
Brief Title: Efficacy of TEAS on Postoperative Pain and Recovery in Patients Undergoing Hepatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024HX1564
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-03

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients who meet the enrollment criteria will be randomized 1:1 to either the transcutaneous electrical acupoint stimulation (TEAS）or the sham groups using a computer-generated random number table. After the randomization, use the opaque envelope, hide each group envelope into an opaque envelope, the envelope outside the code, will be sealed to the researcher, when the study, if the inclusion criteria, then open the corresponding numbered envelope, and intervene according to the group scheme in the envelope.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of participants will be maintained throughout the observation period. The sham group will receive electrode attachment but without stimulation,Throughout the study, for adequate blinding, an opaque tape will be applied to the patient's skin above the electrodes, and the patient's target acupoints will be wrapped in a blanket. All patients will be informed that they might or might not feel a tingling sensation around the acupoints when the TEAS device is working. The patients should not be unblinded until the statistical analysis of the study data is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS group (Experimental): Patients who meet the enrollment criteria will be randomized 1:1 to either the transcutaneous electrical acupoint stimulation (TEAS#or the sham groups. In the TEAS group, the acupoints are bilateral neiguan (PC6) , Hegu(L14), Yanglingquan(GB34), Zusanli(ST 36) and Renying(ST9) acupoints. Patients will receive 30min TEAS before anesthesia until be discharged from the post anaesthesia care unit (PACU). The same treatment for 30 min will be performed on the 1st, 2nd and 3rd days after surgery.The stimulation intensity will be adjusted in accordance with the maximal level tolerated by each patient.
  Interventions: Device: transcutaneous electrical acupoint stimulation
- sham group (Sham Comparator): Patients in the sham group will receive electrode attachment but without stimulation.
  Interventions: Device: sham transcutaneous electrical acupoint stimulation

INTERVENTIONS:
Device: transcutaneous electrical acupoint stimulation — transcutaneous electrical acupoint stimulation Transcutaneous electrical acupoint stimulation (TEAS) is a contemporary modification of traditional acupuncture that sends electrical impulses into acupoints through electrodes on the skin surface. In the TEAS group, patients will receive TEAS 30min before anesthesia until be discharged from the postanaesthesia care unit (PACU). The same treatment will be performed on the 1st, 2nd and 3rd days after surgery.The stimulation intensity will be adjusted in accordance with the maximal level tolerated by each patient.
  Arms: TEAS group
Device: sham transcutaneous electrical acupoint stimulation — Patients in the sham group will receive electrode attachment but without stimulation.
  Arms: sham group

SUMMARY:
The purpose of this study is to access the effect of transcutaneous electrical acupoint stimulation on postoperative pain in patients undergoing hepatectomy

DETAILED DESCRIPTION:
Patients who meet the enrollment criteria will be randomized 1:1 to either the transcutaneous electrical acupoint stimulation (TEAS#or the sham groups. In the TEAS group, the acupoints are bilateral neiguan (PC6) , Hegu(L14), Yanglingquan(GB34), Zusanli(ST 36) and Renying(ST9) acupoints. Patients will receive TEAS 30min before anesthesia until being discharged from the post-anaesthesia care unit (PACU). The same treatment for 30 min will be performed on the 1st, 2nd and 3rd days after surgery.The stimulation intensity will be adjusted in accordance with the maximal level tolerated by each patient.

Patients in the sham group will receive electrode attachment but without stimulation.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80 years old; ASA physical status classⅠ-Ⅲ; Patients scheduled for elective hepatectomy.

Exclusion Criteria:

Have a history of epilepsy; Rash or local infection over the acupoint stimulation skin area; Pregnancy or breastfeeding; Mental retardation, psychiatric, or neurological disease; Inability to comprehend the numeric rating scale (NRS); Implantation of a cardiac pacemaker, cardioverter, or defibrillator; Chronic opioid use; Metastases in other organs;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of moderate to severe pain (NRS ≥ 4) during movement (i.e. cough or take three deep breaths) at 24 hours after surgery | Up to 24 hours postoperatively
  The pain is evaluated using numerical rating scale(NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.

SECONDARY OUTCOMES:
The incidence of moderate to severe pain (NRS ≥ 4) during movement (i.e. cough or take three deep breaths) at 48 and 72 hours after surgery | Up to 72 hours postoperatively
  The pain is evaluated using numerical rating scale(NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.
The incidence of moderate to severe pain (NRS ≥ 4) at rest at 24, 48 and 72 hours after surgery | Up to 72 hours postoperatively
  The pain is evaluated using numerical rating scale(NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.
Pain scores of movement-evoked pain at postoperative 24,48 and 72 hours | Up to 72 hours postoperatively
  The pain is evaluated using numerical rating scale,NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, and 10 points representing the strongest pain.
Pain scores of pain at rest at 24, 48 and 72 hours postoperatively | Up to 72 hours postoperatively
  The pain is evaluated using numerical rating scale,NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, and 10 points representing the strongest pain
The cumulative morphine consumption at 24, 48, and 72 hours postoperatively | Up to 72 hours postoperatively
  Postoperative opioid use is reported as morphine milligram equivalents, calculated using the Practical Pain Management calculator
The incidence of postoperative nausea and vomiting during the first 24,48,72 hours | Up to 72 hours postoperatively
  We considered it PONV if patients felt any nausea or had any vomiting
The incidence of a composite of postoperative pulmonary complications during hospitalization | immediately after the end of surgery, and at the first 24 hours after surgery
  Defined as positive if any component developed before discharge after surgery; These complications included respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, or aspiration pneumonitis loading dose, immediately after the end of surgery, and at the first 24 hours after surgery
Quality of Recovery Scale Score at 24, 48, and 72 hours after surgery | Up to 72 hours postoperatively
  The global QoR-15 score ranges from 0 to 150 and is categorized as five quality of recovery dimensions, including physical comfort (5 items), emotional state (4 items), psychological support (2 items), physical independence (2 items), and pain (2 items). Each piece is graded using an 11-point Likert scale. The QoR is classified according to the QoR-15 score as excellent (QoR-15 > 135), good (122 ≤ QoR-15 ≤ 135), moderate (90 ≤ QoR-15 ≤ 121) and poor (QoR-15 < 90)
Time of Bowel function recovery | Up to 72 hours postoperatively
  Defined as the time to first defecation or time to first flatusdefined as the time to first defecation or time to first flatus defined as the time to first defecation or time to first flatus
Length of hospital stay | From admittance to discharge
  Determined by the number of days from admittance to discharge
The postoperative sleep quality score | Up to 72 hours postoperatively
  Postoperative sleep quality was evaluated using the Athens Insomnia Scale (AIS). The AIS consists of 8 items: waking up at night, sleep induction, final awakening, total sleep duration, sleep quality, well-being, functional ability, and daytime sleepiness. The AIS score ranges from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia.
The anxiety and depression scores | Up to 72 hours postoperatively
  Anxiety and depression score will be evaluated using the Hospital Anxiety and Depression Scale (HADS).The HADS consists of 14 questions, with 7 items each for the anxiety and depression subscales. The score for each item ranges from 0 to 3 points, and scores are summed to yield a separate score for anxiety (HADS-A) and depression (HADS-D).
The incidence of chronic postsurgical pain (CPSP) | 3 months after surgery
  Patients were inquired whether they had any pain （NRS ≥ 1）in surgical area and if the pain developed postoperatively. If subjects answered with a 'no' to any of the two questions, those patients were classified as cases without CPSP. Contrarily, if subjects answered yes, they were considered CPSP cases.

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No